CLINICAL TRIAL: NCT00045760
Title: The Study of Drotrecogin Alfa (Activated) in a Subpopulation of Adult Patients With Severe Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 7252, 6669; F1K-MC-EVCL; F1K-MC-EVCM
Record Dates: First submitted 2002-09-09; First posted 2002-09-10 (Estimated); Last update posted 2006-07-20 (Estimated); Status verified 2006-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — drotrecogin alfa activated

INTERVENTIONS:
Drug: Drotrecogin alfa (activated)

SUMMARY:
Severe sepsis is defined as a systemic inflammatory response syndrome that results from infection and is associated with acute organ dysfunction. It usually results from bacterial infections, but it may occur in response to other pathogens, such as fungi, viruses, and parasites.

DETAILED DESCRIPTION:
Drotrecogin alfa (activated), a recombinant form of human activated protein C, is the first therapeutic intervention shown to reduce all-cause mortality in severe sepsis. In the Phase 3 study (F1K-MC-EVAD; PROWESS), 1690 patients were randomly assigned to receive a 96-hour intravenous infusion of drotrecogin alfa (activated) 24 micrograms/kg/h or placebo (850 patients and 840 patients, respectively). Overall, administration of drotrecogin alfa (activated) yielded a clinically significant reduction in 28-day all-cause mortality: 24.7% of drotrecogin alfa (activated) patients died versus 30.8% of placebo patients (19.4% relative risk reduction; p=0.005; Bernard et al. 2001). The only safety concern noted in the Phase 3 trial was an increased risk of serious bleeding among drotrecogin alfa (activated) patients (3.5% versus 2.0% of placebo patients). The difference between the two treatment groups in the number of patients who experienced a serious bleeding event was due to the greater number of drotrecogin alfa (activated) patients who experienced a serious bleeding event that was related to a procedure (for example, bleeding that resulted from the placement of a catheter or nephrostomy tube). The number of patients who experienced spontaneous serious bleeding events was similar between the two treatment groups.

The Regulatory authorities have approved the use of drotrecogin alfa (activated) in severe sepsis patients with a high level of disease severity and risk of death. Thus, the regulatory authorities have requested a study evaluating drotrecogin alfa (activated) in a specific subpopulation of patients with severe sepsis and at lower risk of death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with severe sepsis.
* Presence of a suspected or proven infection.
* One or more sepsis-associated organ failure.

Exclusion Criteria:

* Are indicated for the treatment with drotrecogin alfa (activated) in the investigative site country.
* Are contraindicated for treatment with drotrecogin alfa (activated) under the applicable label in the investigative site country.
* Platelet count <30,000/mm3.
* Are receiving therapeutic heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Locations (426):
- United States (152):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tuscon, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Berkeley, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Fullerton, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santa Barbara, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Englewood, Colorado
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Loveland, Colorado
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Milford, Connecticut
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Stamford, Connecticut
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brandon, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lakeland, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sarasota, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Weston, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Albany, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Austell, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Riverdale, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Berwyn, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Decatur, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Elk Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Oak Park, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New Albany, Indiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Olathe, Kansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Crestview Hills, Kentucky
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Covington, Louisiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Portland, Maine
  - timoreFor additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Barrien Springs, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Royal Oak, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ypsilanti, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saint Paul, Minnesota
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., City of Saint Peters, Missouri
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Missoula, Montana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hackensack, New Jersey
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Neptune City, New Jersey
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Phillipsburg, New Jersey
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., East Meadow, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Johnson City, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Larchmont, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Manhasset, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New Hyde Park, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hendersonville, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bismarck, North Dakota
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Manfield, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Youngstown, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Abington, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., East Stroudsburg, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Erie, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jefferson Hills, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Reading, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sayre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., York, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Chattanoga, Tennessee
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jackson, Tennessee
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., El Paso, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Fort Sam Houston, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Forth Worth, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Galveston, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Irving, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lackland Air Force Base, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Odessa, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Alexandria, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lynchburg, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Huntington, West Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Morgantown, West Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Milwaukee, Wisconsin
- Australia (21):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Camperdown, New South Wales
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kingswood, New South Wales
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Liverpool, New South Wales
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Randwick, New South Wales
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tiwi, Northern Territory
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Douglas, Queensland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Herston, Queensland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Adelaide, South Australia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bedford Park, South Australia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hobart, Tasmania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Dandenong, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Fitzroy, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Footscray, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Heidelberg, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Parkville, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Prahran, Victoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nedlands, Western Australia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Perth, Western Australia
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Innsbruck, Innsbruck
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vienna, Vienna
- Belgium (7):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brussells, Brussells
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brussels, Brussels Capital
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ghent, Gent
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Liège, Liege
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mons, Mons
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ottignies, Ottignies
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Yvior, Yvior
- Brazil (9):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Salvador, Estado de Bahia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Curitiba, Paraná
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Porto Alegre, Porto Alegre
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rio de Janeiro, Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Rio de Janeiro, Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Florianópolis, Santa Catarina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., São Paulo, São Paulo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., São Paulo, São Paulo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Porto Alegre
- Canada (20):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New Westminster, British Columbia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saint John, New Brunswick
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brampton, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Windsor, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Greenfield Park, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sherbrooke, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Regina, Saskatchewan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saskatoon, Saskatchewan
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Independencia, Santiago Metropolitan, Chile
- Czechia (9):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Brno, Brno
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hradec Králové, Hradec Kralove
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Olomouc, Olomouc
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ostrava Poruba, Ostrava Poruba
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pilsen, Plzen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Prague, Praha 10
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Prague, Praha 2
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Praha 5 Motol, Praha 5 Motol
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Prague, Praha 8
- Denmark (4):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Esbjerg, Esbjerg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hvidovre, Hvidovre
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Roskilde, Roskilde
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Viborg, Viborg
- Egypt (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cairo, Cairo Governorate
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Alexandria
- Finland (6):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Helsinki, Hus, Helsinki, Hus
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jyväskylä, Jyvaskyla
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Kuopio, Kuopio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Oulu, Oulu
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician, Turku, Turku
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Tampere
- France (35):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Argenteuil, Argenteuil
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Aulnay-sous-Bois, Aulnay-Sous-Bois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Besançon, Besancon Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bondy, Bondy Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Clichy, Clichy
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Corbeil-Essonnes, Corbeil Essonnes Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Dijon, Dijon Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Gleizé, Gleize
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Le Chesnay, Le Chesnay Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Le Kremlin-Bicêtre, Le Kremlin Bicetre Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lille, Lille Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lille, Lille
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Limoges, Limoges Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lyon, Lyon Cedex 03
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Marseille, Marseille Cedex 09
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nancy, Nancy
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nice, Nice Cedex 1
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nice, Nice Cedex 3
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nîmes, Nimes
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Orléans, Orleans Cedex 2
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Paris, Paris Cedex 10
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Paris, Paris Cedex 13
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Paris, Paris Cedex 14
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Poissy, Poissy
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Poitiers, Poitiers
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pontoise, Pontoise Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saint-Denis, Saint Denis Cedex 1
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saint-Etienne, Saint Etienne Cedex 2
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Strasbourg, Strasbourg Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Toulouse, Toulouse
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tours, Tours Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vesoul, Vesoul
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Garches
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Longsumeau Cedex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Rennes
- Germany (18):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Aachen, Aachen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bonn, Bonn
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bremen, City state Bremen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Erfurt, Erfurt
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Freiburg im Breisgau, Freiburg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Halle, Halle
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hamburg, Hamburg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hanover, Hannover
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Essen, Hesse
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Leipzig, Leipzig
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lübeck, Lubeck
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mannheim, Mannheim
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., München, Munchen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Regensburg, Regensburg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Reutlingen, Reutlingen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Berlin, State of Berlin
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tübingen, Tubingen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Göttingen
- India (7):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hyderabad, Andhara Pradesh
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hyderabad, Hyderabad
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bangalore, Karnataka
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mumbai, Maharashtra
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pune, Maharashtra
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., New Delhi, National Capital Territory of Delhi
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Noida, Uttar Pradesh
- Italy (32):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ancona, Ancona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Arezzo, Arezzo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Carbonara, Bari
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bergamo, Bergamo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bologna, Bologna
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bolzano, Bolzano
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cagliari, Cagliari
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Como, Como
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Catania, CT
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ferrara, Ferrara
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lecce, Lecce
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lecco, Lecco
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Milan, Milano
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vimercate, Milano
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Monza, MI
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Padua, Padova
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Palermo, Palermo
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pavia, Pavia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Pordenone, PD
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pesaro, Pesaro
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pisa, Pisa
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Roma, roma
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sassari, sassari
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pietra Ligure, Savona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Siena, Siena
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Treviglio, Treviglio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Trieste, Trieste
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Varese, Varese
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Arzignano, Vicenza
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vicenza, Vicenza
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Palermo
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Beirut, Beyrouth, Lebanon
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Mexico City, Mexico City
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Monterrey, Nuevo León
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Apeldoorn, Apeldoorn
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Breda, Breda
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., 's-Hertogenbosch, Den Bosch
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tilburg, Tilburg
- New Zealand (4):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Auckland, Auckland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Christchurch, Canterbury
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hamilton, Hamilton
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hastings, Hastings
- Norway (5):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ålesund, Alesund
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Drammen, Drammen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nordbyhagen, Nordbyhagen
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Oslo, Oslo County
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Trondheim, Trondheim
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bucharest, Bucharest
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bucharest, Sector 2
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Moscow, Russia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saint Peterburg, Russia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Smolensk, Smolensk Oblast
- Saudi Arabia (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jeddah, Jeddah
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Riyadh, Riyadh Region
- For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Singapore, Singapore
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bratislava, Bratislava Region
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Košice, Košice Region
- South Africa (7):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bloemfontein, Bloemfontein
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Somerset West, Cape Province
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Kimberley, Northern Cape
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Pretoria, Pretoria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Thaba Tshwane, Thaba Tshwane
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Medunsa
- Spain (27):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Alicante, Alicante
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., San Juan, Alicante
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Badajoz, Badajoz
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Barcelona, Barcelona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Girona, Barcelona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sabadell, Barcelona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Burgos, Burgos
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cadiz, Cadiz
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Jerez de la Frontera, Cadiz
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santander, Cantabria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Castellon, Castellon
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Las Palmas, Gran Canaria
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santiago Compostela, La Coruna
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Alcorcón, Madrid
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Getafe, Madrid
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Leganés, Madrid
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Madrid, Madrid
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Murcia, Murcia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Palencia, Palencia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Palma de Mallorca, Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Salmanca, Salmanca
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Santa Cruz de Tenerife, Santa Cruz De Tenerife
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Seville, Sevilla
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Valencia, Valencia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Valladolid, Valladolid
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Galdakao, Vizcaya
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Terrassa
- Sweden (9):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Falun, Falun
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Gothenburg, Goteborg
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Huddinge, Huddinge
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kristianstad, Kristianstad
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Östersund, Ostersund
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Stockholm, Stockholm County
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sundsvall, Sundsvall
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Karistad
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Skövde
- Switzerland (3):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bern, Canton of Bern
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Zurich, Canton of Zurich
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Geneva
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Neihu Taipei, R. O. C.
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Taipei
- Thailand (2):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Bangkok
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Khon Kaen
- United Kingdom (25):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Bradford, Bradford
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cardiff, Cardiff
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Plymouth, Devon
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Langside, Glasgow
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Portsmouth, Hampshire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Royal Tunbridge Wells, Kent
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Manchester, Lancashire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Leicester, Leicestershire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Reading, London Road
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., London, London
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., London, London
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Waterloo, London
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Wythenshawe, Manchester
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Harrow, Middlesex
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kings Lynn, Norfolk
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Norwich, Norfolk
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Northampton, Northampton
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Nottingham, Nottinghamshire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Aberdeen, Scotland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Livingstone, West Lothian
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Birmingham, West Midlands
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Leeds, West Yorkshire